CLINICAL TRIAL: NCT00065858
Title: A Randomized, Controlled Trial of the Efficacy, Safety, and Acceptability of BufferGel
Brief Title: Effectiveness of BufferGel as a Vaginal Contraceptive
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Premier Research (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CCN003; NCT00397618 (obsolete NCT alias)
Record Dates: First submitted 2003-08-01; First posted 2003-08-05 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Pregnancy
Keywords: Contraception; Nonoxynol 9; Microbicide; Spermicide
MeSH Terms: interventions — BufferGel

INTERVENTIONS:
Drug: BufferGel

SUMMARY:
BufferGel is a new contraceptive gel designed to be used with a diaphragm. In addition to preventing pregnancy, BufferGel may also prevent some types of sexually transmitted diseases (STDs). This study will compare BufferGel to Gynol II, a currently available contraceptive gel.

DETAILED DESCRIPTION:
Vaginal acidity is thought to be one means by which the vagina prevents overgrowth or colonization by harmful microbial flora. Sperm and many STD pathogens, including HSV-1 and HSV-2, Neisseria gonorrhoeae, Treponema pallidum, Haemophilus ducreyi, and a variety of bacterial vaginosis-associated bacteria, are inactivated at pH less than 5 in vitro. BufferGel, a vaginal spermicide and microbicide, is an acidic buffer that maintains the vagina at or near its natural state of mild acidity. Formulated at vaginal pH (pH 3.9), BufferGel prevents or limits the semen-induced rise in vaginal pH. Carbopol 974P, the buffering agent in BufferGel, is a high molecular weight, cross-linked, polyacrylic acid used as a gelling or tableting agent in many pharmaceuticals; it has a well-documented record of mucosal safety in animals and humans. This study will determine the safety and contraceptive efficacy of BufferGel spermicide used with a diaphragm compared to Gynol II spermicide used with a diaphragm. The study will also measure the frequency of bacterial vaginosis, urinary tract infections, and cervical lesions in women using BufferGel compared with Gynol II.

Participants in this study will be fitted for a diaphragm and randomized to receive either BufferGel or Gynol II. All participants will be instructed on the use of the test product with the diaphragm. Participants will be followed through 6 menstrual cycles (approximately 7 months) and will have 4 study visits and one study phone call. Some participants may enroll in an extended version of the study and be followed for an additional 6 cycles and 2 additional study visits. Study visits will include a gynecologic exam, Pap smear, and blood and urine tests. Participants will be asked to keep a diary to record information on product use. Some participants may also be asked to enroll in a colposcopy substudy. These participants will undergo colposcopy at study entry and after cycles 1, 3 and 6.

ELIGIBILITY:
Inclusion Criteria

* General good health
* Sexually active, at risk for pregnancy, and desiring contraception
* Low-risk for HIV or STD infection
* Single sexual partner who is at low-risk for HIV or STD infection for 6 months prior to study entry
* Expect to have same sexual partner for duration of the study
* Normal cyclic menses with a usual length of 21 to 35 days
* Documented history of at least two spontaneous, normal menstrual cycles since delivery, abortion, or after discontinuing hormonal contraception/hormonal therapy
* Willing to accept a risk of pregnancy
* Willing to engage in an average of 1 to 2 acts of heterosexual vaginal intercourse per week for a period of 6 months
* Willing to be fitted with a diaphragm and use the diaphragm with test product during all acts of heterosexual vaginal intercourse for the duration of the study
* Willing to only use the test product with diaphragm as the sole method of contraception over the course of the study (with the exception of emergency contraceptive pills when indicated)
* Capable of using the product and diaphragm properly
* Willing to keep a diary to record coital information, product use information, information about the use of other vaginal products, and sign and symptom data for self and partner
* Agree not to participate in any other clinical trials during the course of the study
* Written informed consent to participate in the trial

Participant's Sexual Partner Must Not Be/Have

* Infertile
* Treated for Chlamydia trachomatis or Neisseria gonorrhoeae in the 6 months prior to study entry
* HIV infected
* More than one sexual partner in the 4 months prior to study entry
* Engaged in homosexual intercourse
* Shared injection drug needles in the 6 months prior to study entry
* Allergy or sensitivity to spermicides or products containing Nonoxynol 9 or latex

Exclusion Criteria

* Pregnant or desire to become pregnant during the course of the study
* History of infertility or conditions that may lead to infertility
* Allergy or sensitivity to spermicides or products containing Nonoxynol 9 or latex
* History of toxic shock syndrome (TSS)
* Two or more urinary tract infections (UTIs) in the 12 months prior to study entry
* Current suspected or diagnosed urinary tract infection or vaginitis
* Contraindications to pregnancy (medical condition or chronic use of medications contraindicated for pregnancy)
* Treated with antibiotics for pelvic inflammatory disease (PID) without a subsequent intrauterine pregnancy
* More than one sexual partner in the 4 months prior to study entry
* Shared injection drug needles in the 6 months prior to study entry
* HIV infected or suspected HIV infection
* Genital herpes simplex virus (HSV) infection with the first occurrence (initial episode) within 3 months prior to study entry or have clinical evidence of HSV on exam
* Sexually transmitted diseases (STDs) in the 3 months prior to study entry
* Lactating or breastfeeding
* Abnormal vaginal bleeding or spotting in the month prior to study entry
* Lower abdominal or pelvic pain in the month prior to study entry
* Abnormal finding on pelvic examination which, in the view of the study investigator, precludes participation in study
* Vaginal or cervical irritation, including vaginal or cervical epithelial disruption, ulceration, bleeding, petechiae, sloughing, or areas of obvious erythema
* Vaginal or cervical biopsy or surgery in the 3 months prior to study entry
* Vaginal or systemic antibiotics, antivirals, or antifungals in the 14 days prior to study entry
* Depo-Provera injection in the 10 months prior to study
* Vaginal or cervical abnormality that would interfere with the proper placement and retention of test product and diaphragm
* Abnormal Pap smear in the 12 months prior to study entry
* Consume (on average) greater than 2 to 3 alcoholic beverages per day
* Drug abuse (recreational, prescription, or OTC) in the 12 months prior to study entry
* Investigational drug or device use in the month prior to study entry
* Previously participated in or completed this study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 975
Dates: Start 2001-09; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Overall Officials: H. Trent MacKay, MD, MPH, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (9):
- United States (9):
  - California Family Health Council, Berkeley, California
  - California Family Health Council, Los Angeles, California
  - University of Colorado, Denver, Colorado
  - New York University, New York, New York
  - Columbia University, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Eastern Virginia Medical School, Norfolk, Virginia

REFERENCES:
- [Derived] Barnhart KT, Rosenberg MJ, MacKay HT, Blithe DL, Higgins J, Walsh T, Wan L, Thomas M, Creinin MD, Westhoff C, Schlaff W, Archer DF, Ayers C, Kaunitz A, Das S, Moench TR. Contraceptive efficacy of a novel spermicidal microbicide used with a diaphragm: a randomized controlled trial. Obstet Gynecol. 2007 Sep;110(3):577-86. doi: 10.1097/01.AOG.0000278078.45640.13. PMID 17766603